CLINICAL TRIAL: NCT02070380
Title: Phase IV, Double Blind, Multi-Center, Randomized, Two-Arm Crossover Study to Compare 0.1 mmol/kg of MultiHance With 0.1 mmol/kg of Dotarem and 0.05 mmol/kg of MultiHance With 0.1 mmol/kg of Dotarem in MRI of the Brain
Brief Title: Crossover Comparison of MultiHance and Dotarem
Acronym: BENEFIT
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Bracco Diagnostics, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Diagnostic
Other Study IDs: MH-148
Record Dates: First submitted 2014-02-20; First posted 2014-02-25 (Estimated); Results first posted 2017-01-10 (Estimated); Last update posted 2017-01-10 (Estimated); Status verified 2016-11

CONDITIONS: Brain Disease
Keywords: confirmed brain disease; highly suspected brain disease
MeSH Terms: conditions — Brain Diseases | interventions — gadobenic acid; gadoterate meglumine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- MultiHance 0.1 then Dotarem 0.1 mmol/kg (Experimental): MultiHance 0.1 mmol/kg Then Dotarem 0.1 mmol/kg
  Interventions: Drug: MultiHance 0.1 mmol/kg; Drug: Dotarem
- MultiHance 0.05 then Dotarem 0.1 mmol/kg (Experimental): MultiHance 0.05 mmol/kg Then Dotarem 0.1 mmol/kg
  Interventions: Drug: Dotarem; Drug: MultiHance 0.05 mmol/kg
- Dotarem 0.1 then MultiHance 0.1 mmol/kg (Active Comparator): Dotarem 0.1 mmol/kg Then MultiHance 0.1 mmol/kg
  Interventions: Drug: MultiHance 0.1 mmol/kg; Drug: Dotarem
- Dotarem 0.1 then MultiHance 0.05 mmol/kg (Active Comparator): Dotarem 0.1 mmol/kg Then MultiHance 0.05 mmol/kg
  Interventions: Drug: Dotarem; Drug: MultiHance 0.05 mmol/kg

INTERVENTIONS:
Drug: MultiHance 0.1 mmol/kg — MultiHance administered at 0.1 mmol/kg
  Arms: Dotarem 0.1 then MultiHance 0.1 mmol/kg; MultiHance 0.1 then Dotarem 0.1 mmol/kg
Drug: Dotarem — Dotarem administered at 0.1 mmol/kg
  Other Names: Dotarem 0.1 mmol/kg
Drug: MultiHance 0.05 mmol/kg — MultiHance administered at 0.05 mmol/kg
  Arms: Dotarem 0.1 then MultiHance 0.05 mmol/kg; MultiHance 0.05 then Dotarem 0.1 mmol/kg

SUMMARY:
This study aims at a comparison between MultiHance at a dose of 0.1 mmol/kg and 0.05 mmol/kg and Dotarem at a dose of 0.1 mmol/kg in brain tumor patients to show superiority of MultiHance.

DETAILED DESCRIPTION:
This crossover study aims at a comparison between 0.1 mmol/kg MultiHance and 0.1 mmol/kg Dotarem, between 0.05 MultiHance and 0.1 mmol/kg Dotarem in terms of diagnostic preference at CE-MRI in brain tumor patients to show superiority of MultiHance.

ELIGIBILITY:
Inclusion Criteria:

* Are at least 18 years of age or older
* Are able to give written informed consent and are willing to comply with the protocol requirements
* Are scheduled to undergo MRI
* Are willing to undergo two MRI procedures within 14 days
* Have confirmed or are highly suspected to have brain tumor(s) (primary or secondary), as determined by:
* Clinical/neurological symptomatology;
* Diagnostic testing, such as CT or previous MRI examinations; or
* Have had recent brain surgery and are to be evaluated for recurrence

Exclusion Criteria:

* Are pregnant or lactating females. Exclude the possibility of pregnancy:
* By testing on site at the institution within 24 hours prior to the start of each investigational product administration; or
* By history (i.e., tubal ligation or hysterectomy); or
* Post menopausal with a minimum of 1 year without menses
* Have any known allergy to one or more of the ingredients in the investigational products, or have a history of hypersensitivity to any metals
* Have congestive heart failure (class IV according to the classification of the New York Heart Association)
* Have suffered a stroke within a year
* Have received or are scheduled to receive any other contrast medium in the 24 hours preceding through the 24 hours following Exam 1, and in the 24 hours preceding through the 24 hours following Exam 2
* Have received or are scheduled to receive an investigational compound and/or medical device within 30 days before admission into the present study, through the 24 hours post-administration of the second investigational product
* Have moderate-to-severe renal impairment, defined as Glomerular Filtration Rate (GFR)/estimated GFR < 45 mL/min
* Have been previously entered into this study
* Have received or are scheduled for one of the following:
* Surgical or chemotherapeutic treatment within three weeks prior to the first examination or between the two examinations
* Initiation of steroid therapy between the two examinations
* Radiosurgery between the two examinations
* Have any contraindications to MRI such as a pace-maker, magnetic material (i.e., surgical clips) or any other conditions that would preclude proximity to a strong magnetic field
* Are suffering from severe claustrophobia
* Have any medical condition or other circumstances which would significantly decrease the chances of obtaining reliable data, achieving study objectives, or completing the study and/or post-dose follow-up examinations

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 179 (Actual)
Dates: Start 2014-02; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gianpaolo Pirovano, MD, Study Director — Bracco Diagnostics, Inc
Locations (1):
- Samaritan Health Services, Corvallis, Oregon, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 179 patients were recruited from February 2014 through February 2015 at 14 clinical trial sites. Off-site assessment of the images was performed between 19 February - 17 March 2015 by 3 board-certified neuroradiologists blinded as to which contrast agent was used, patient clinical information, and the results of other imaging studies.
Pre-assignment Details: 179 patients were enrolled and signed informed consent. Each enrolled patient was randomized and 177 were dosed with at least one contrast agent.
Groups:
- MultiHance 0.1 mmol/kg Then Dotarem 0.1 mmol/kg: Patients randomized to receive MultiHance 0.1 mmol/kg first
- Dotarem 0.1 mmol/kg Then MultiHance 0.1 mmol/kg; Dotarem 0.1 mmol/kg Then MultiHance 0.05 mmol/kg: Patients randomized to receive Dotarem 0.1 mmol/kg first
- MultiHance 0.05 mmol/kg Then Dotarem 0.1 mmol/kg: Patients randomized to receive MultiHance 0.05 mmol/kg first
Period: First Injection
Arm/Group | MultiHance 0.1 mmol/kg Then Dotarem 0.1 mmol/kg | Dotarem 0.1 mmol/kg Then MultiHance 0.1 mmol/kg | MultiHance 0.05 mmol/kg Then Dotarem 0.1 mmol/kg | Dotarem 0.1 mmol/kg Then MultiHance 0.05 mmol/kg
Started | 31 | 39 | 53 | 54
Completed | 31 | 39 | 53 | 54
Not Completed | 0 | 0 | 0 | 0
Period: Washout (no Second Injection/MRI)
Arm/Group | MultiHance 0.1 mmol/kg Then Dotarem 0.1 mmol/kg | Dotarem 0.1 mmol/kg Then MultiHance 0.1 mmol/kg | MultiHance 0.05 mmol/kg Then Dotarem 0.1 mmol/kg | Dotarem 0.1 mmol/kg Then MultiHance 0.05 mmol/kg
Started | 31 | 39 | 53 | 54
Completed | 31 | 34 | 51 | 51
Not Completed | 0 | 5 | 2 | 3
Not completed — Withdrawal by Subject | 0 | 5 | 2 | 3
Period: Second Injection
Arm/Group | MultiHance 0.1 mmol/kg Then Dotarem 0.1 mmol/kg | Dotarem 0.1 mmol/kg Then MultiHance 0.1 mmol/kg | MultiHance 0.05 mmol/kg Then Dotarem 0.1 mmol/kg | Dotarem 0.1 mmol/kg Then MultiHance 0.05 mmol/kg
Started | 31 | 34 | 51 | 51
Completed | 31 | 32 | 50 | 46
Not Completed | 0 | 2 | 1 | 5
Not completed — Image sets missing or technically inadeq | 0 | 1 | 0 | 0
Not completed — Protocol Violation | 0 | 1 | 1 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | MultiHance 0.1 mmol/kg Then Dotarem 0.1 mmol/kg | Dotarem 0.1 mmol/kg Then MultiHance 0.1 mmol/kg | MultiHance 0.05 mmol/kg Then Dotarem 0.1 mmol/kg | Dotarem 0.1 mmol/kg Then MultiHance 0.05 mmol/kg | Total
Number analyzed (Participants) | 31 | 32 | 50 | 46 | 159
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 24 | 20 | 36 | 28 | 108
  >=65 years | 7 | 12 | 14 | 18 | 51
Gender [Count of Participants; unit: Participants]
  Female | 20 | 20 | 25 | 22 | 87
  Male | 11 | 12 | 25 | 24 | 72
Race/Ethnicity, Customized [Number; unit: participants]
  White | 31 | 31 | 46 | 46 | 154
  Black | 0 | 1 | 2 | 0 | 3
  Asian | 0 | 0 | 1 | 0 | 1
  Other | 0 | 0 | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 12 | 15 | 21 | 21 | 69
  Europe | 19 | 17 | 29 | 25 | 90

OUTCOME MEASURES:

1. Primary Outcome: Global Diagnostic Preference Between the Two Exams
Description: Assessed by 3 blinded readers for each of the 159 patients who had post-dose exams for both MultiHance, 0.1 mmol/kg and 0.05 mmol/kg doses, and Dotarem 0.1 mmol/kg. Readers assessed whether images with MultiHance were preferred or images with Dotarem were preferred, or whether images after both exams were considered equal. An image set deemed technically inadequate by a blinded reader was excluded from efficacy analysis for that specific reader. Therefore, the number of participant exams evaluated by each reader differed slightly across readers and endpoints.
Time Frame: Comparison of image sets obtained within 2 to 14 days
Population: Per Protocol=patients who completed both exams, had global paired image data available, and had no major protocol violations
Measure: Number; unit: participant exams
Groups:
- MultiHance 0.1 mmol/kg Arm (Reader 1); MultiHance 0.1 mmol/kg Arm (Reader 2); MultiHance 0.1 mmol/kg Arm (Reader 3): MRI with MultiHance 0.1 mmol/kg versus MRI with Dotarem 0.1 mmol/kg
- MultiHance 0.05 mmol/kg Arm (Reader 1); MultiHance 0.05 mmol/kg Arm (Reader 2); MultiHance 0.05 mmol/kg Arm (Reader 3): MRI with MultiHance 0.05 mmol/kg versus MRI with Dotarem 0.1 mmol/kg
Arm/Group | MultiHance 0.1 mmol/kg Arm (Reader 1) | MultiHance 0.1 mmol/kg Arm (Reader 2) | MultiHance 0.1 mmol/kg Arm (Reader 3) | MultiHance 0.05 mmol/kg Arm (Reader 1) | MultiHance 0.05 mmol/kg Arm (Reader 2) | MultiHance 0.05 mmol/kg Arm (Reader 3)
Number analyzed (Participants) | 63 | 62 | 62 | 96 | 94 | 95
participant exams
  MultiHance Preferred | 31 | 51 | 43 | 14 | 18 | 15
  Contrast Agents Equal | 31 | 9 | 17 | 75 | 56 | 63
  Dotarem Preferred | 1 | 2 | 2 | 7 | 20 | 17
Statistical Analysis 1: Comparison: MultiHance 0.1 mmol/kg Arm (Reader 1); Null hypotheses: A 0.1 mmol/kg dose of MULTIHANCE is equal to a 0.1 mmol/kg dose of DOTAREM, in terms of the assessment of global diagnostic preference in an off-site pre-dose plus postdose paired global assessment; Test type: Superiority or Other; p < 0.0001, Wilcoxon signed-rank test. — Only 1 primary endpoint, no adjustment for multiple comparisons and the a priori threshold for statistical significance was 0.05; ∆Percentage MH better minus DM better = 47.6, 95% CI 2-sided [34.5 to 60.7] — Difference in percentage MultiHance better minus percentage Dotarem better (%) , 2-sided 95% confidence interval was estimated using Altman's general approximate normal method
Statistical Analysis 2: Comparison: MultiHance 0.05 mmol/kg Arm (Reader 1); Null hypotheses: A 0.05 mmol/kg dose of MULTIHANCE is equal to a 0.1 mmol/kg dose of DOTAREM, in terms of the assessment of global diagnostic preference in an off-site pre-dose plus post-dose paired global assessment; Test type: Superiority or Other; p = 0.1295, Wilcoxon signed-rank test. — [p-value comment as in outcome 1, analysis 1]; ∆Percentage MH better minus DM better = 7.3, 95% CI 2-sided [-2.0 to 16.5] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: MultiHance 0.1 mmol/kg Arm (Reader 2); [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.0001, Wilcoxon signed rank test — [p-value comment as in outcome 1, analysis 1]; ∆Percentage MH better minus DM better = 79.0, 95% CI 2-sided [67.1 to 91.0] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 4: Comparison: MultiHance 0.05 mmol/kg Arm (Reader 2); [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.7503, Wilcoxon signed rank test — [p-value comment as in outcome 1, analysis 1]; Percentage MH better minus DM better = -2.1, 95% CI 2-sided [-15.0 to 10.7] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 5: Comparison: MultiHance 0.1 mmol/kg Arm (Reader 3); Null hypotheses: A 0.1 mmol/kg dose of MULTIHANCE is equal to a 0.1 mmol/kg dose of DOTAREM, in terms of the assessment of global diagnostic preference in an off-site pre-dose plus post-dose paired global assessment; Test type: Superiority or Other; p < 0.0001, Wilcoxon signed rank test — [p-value comment as in outcome 1, analysis 1]; ∆Percentage MH better minus DM better = 66.1, 95% CI 2-sided [52.8 to 79.5] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 6: Comparison: MultiHance 0.05 mmol/kg Arm (Reader 3); [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.7297, Wilcoxon signed rank test — [p-value comment as in outcome 1, analysis 1]; ∆Percentage MH better minus DM better = -2.1, 95% CI 2-sided [-13.8 to 9.6] — [estimate comment as in outcome 1, analysis 1]

2. Secondary Outcome: Lesion Border Delineation
Description: as for outcome 1
Time Frame: Comparison of image sets obtained within 2 to 14 days
Measure: Number; unit: participant exams
Arm/Group | MultiHance 0.1 mmol/kg Arm (Reader 1) | MultiHance 0.1 mmol/kg Arm (Reader 2) | MultiHance 0.1 mmol/kg Arm (Reader 3) | MultiHance 0.05 mmol/kg Arm (Reader 1) | MultiHance 0.05 mmol/kg Arm (Reader 2) | MultiHance 0.05 mmol/kg Arm (Reader 3)
Number analyzed (Participants) | 63 | 62 | 62 | 96 | 94 | 95
participant exams
  MultiHance Preferred | 29 | 34 | 25 | 11 | 12 | 8
  Contrast Agents Equal | 33 | 27 | 35 | 76 | 66 | 77
  Dotarem Preferred | 1 | 1 | 2 | 9 | 16 | 10
Statistical Analysis 1: Comparison: MultiHance 0.1 mmol/kg Arm (Reader 1); This is a secondary analysis. Null hypotheses: A 0.1 mmol/kg dose of MULTIHANCE is equal to a 0.1 mmol/kg dose of DOTAREM, in terms of the assessment of Lesion Border Delineation in an off-site pre-dose plus postdose paired global assessment; Test type: Superiority or Other; p < 0.0001, Wilcoxon signed-rank test — The priori threshold for statistical significance was 0.05
Statistical Analysis 2: Comparison: MultiHance 0.05 mmol/kg Arm (Reader 1); This is a secondary analysis. Null hypotheses: A 0.05 mmol/kg dose of MULTIHANCE is equal to a 0.1 mmol/kg dose of DOTAREM, in terms of the assessment of Lesion Border Delineation in an off-site pre-dose plus post-dose paired global assessment; Test type: Superiority or Other; p = 0.8238, Wilcoxon signed-rank test — The priori threshold for statistical significance was 0.05
Statistical Analysis 3: Comparison: MultiHance 0.1 mmol/kg Arm (Reader 2); [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p < 0.0001, Wilcoxon signed rank test — The priori threshold for statistical significance was 0.05
Statistical Analysis 4: Comparison: MultiHance 0.05 mmol/kg Arm (Reader 2); This is a secondary analysis. Null hypotheses: A 0.05 mmol/kg dose of MULTIHANCE is equal to a 0.1 mmol/kg dose of DOTAREM, in terms of the assessment of Lesion Border Delineation in an off-site pre-dose plus postdose paired global assessment; Test type: Superiority or Other; p = 0.4597, Wilcoxon signed rank test — The priori threshold for statistical significance was 0.05
Statistical Analysis 5: Comparison: MultiHance 0.1 mmol/kg Arm (Reader 3); [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p < 0.0001, Wilcoxon signed rank test — The priori threshold for statistical significance was 0.05
Statistical Analysis 6: Comparison: MultiHance 0.05 mmol/kg Arm (Reader 3); [analysis description as in outcome 2, analysis 4]; Test type: Superiority or Other; p = 0.8145, Wilcoxon signed rank test — The priori threshold for statistical significance was 0.05

3. Secondary Outcome: Lesion Internal Morphology
Description: as for outcome 1
Time Frame: Comparison of image sets obtained within 2 to 14 days
Measure: Number; unit: participant exams
Arm/Group | MultiHance 0.1 mmol/kg Arm (Reader 1) | MultiHance 0.1 mmol/kg Arm (Reader 2) | MultiHance 0.1 mmol/kg Arm (Reader 3) | MultiHance 0.05 mmol/kg Arm (Reader 1) | MultiHance 0.05 mmol/kg Arm (Reader 2) | MultiHance 0.05 mmol/kg Arm (Reader 3)
Number analyzed (Participants) | 63 | 62 | 62 | 96 | 94 | 95
participant exams
  MultiHance better | 10 | 14 | 23 | 4 | 3 | 5
  No Difference Between MultiHance and Dotarem | 53 | 48 | 38 | 88 | 87 | 82
  Dotarem better | 0 | 0 | 1 | 4 | 4 | 8
Statistical Analysis 1: Comparison: MultiHance 0.1 mmol/kg Arm (Reader 1); Null hypotheses: A 0.1 mmol/kg dose of MULTIHANCE is equal to a 0.1 mmol/kg dose of DOTAREM, in terms of the assessment of Lesion Internal Morphology in an off-site pre-dose plus postdose paired global assessment; Test type: Superiority or Other; p = 0.0020, Wilcoxon signed-rank test
Statistical Analysis 2: Comparison: MultiHance 0.05 mmol/kg Arm (Reader 1); Null hypotheses: A 0.05 mmol/kg dose of MULTIHANCE is equal to a 0.1 mmol/kg dose of DOTAREM, in terms of the assessment of Lesion Internal Morphology in an off-site pre-dose plus post-dose paired global assessment; Test type: Superiority or Other; p = 1.0000, Wilcoxon signed-rank test
Statistical Analysis 3: Comparison: MultiHance 0.1 mmol/kg Arm (Reader 2); [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.0001, Wilcoxon signed-rank test
Statistical Analysis 4: Comparison: MultiHance 0.05 mmol/kg Arm (Reader 2); Null hypotheses: A 0.05 mmol/kg dose of MULTIHANCE is equal to a 0.1 mmol/kg dose of DOTAREM, in terms of the assessment of Lesion Internal Morphology in an off-site pre-dose plus postdose paired global assessment; Test type: Superiority or Other; p = 1.0000, Wilcoxon signed-rank test
Statistical Analysis 5: Comparison: MultiHance 0.1 mmol/kg Arm (Reader 3); [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p < 0.0001, Wilcoxon signed-rank test
Statistical Analysis 6: Comparison: MultiHance 0.05 mmol/kg Arm (Reader 3); [analysis description as in outcome 3, analysis 4]; Test type: Superiority or Other; p = 0.5811, Wilcoxon signed-rank test

4. Secondary Outcome: Extent of Disease
Description: as for outcome 1
Time Frame: Comparison of image sets obtained within 2 to 14 days
Measure: Number; unit: participant exams
Arm/Group | MultiHance 0.1 mmol/kg Arm (Reader 1) | MultiHance 0.1 mmol/kg Arm (Reader 2) | MultiHance 0.1 mmol/kg Arm (Reader 3) | MultiHance 0.05 mmol/kg Arm (Reader 1) | MultiHance 0.05 mmol/kg Arm (Reader 2) | MultiHance 0.05 mmol/kg Arm (Reader 3)
Number analyzed (Participants) | 63 | 62 | 62 | 96 | 94 | 95
participant exams
  MultiHance Better | 15 | 18 | 15 | 6 | 5 | 7
  No Difference between MultiHance and Dotarem | 48 | 43 | 45 | 84 | 83 | 80
  Dotarem Better | 0 | 1 | 2 | 6 | 6 | 8
Statistical Analysis 1: Comparison: MultiHance 0.1 mmol/kg Arm (Reader 1); Null hypotheses: A 0.1 mmol/kg dose of MULTIHANCE is equal to a 0.1 mmol/kg dose of DOTAREM, in terms of the assessment of Extent of Disease in an off-site pre-dose plus postdose paired global assessment; Test type: Superiority or Other; p < 0.0001, Wilcoxon signed-rank test
Statistical Analysis 2: Comparison: MultiHance 0.05 mmol/kg Arm (Reader 1); Null hypotheses: A 0.05 mmol/kg dose of MULTIHANCE is equal to a 0.1 mmol/kg dose of DOTAREM, in terms of the assessment of Extent of Disease in an off-site pre-dose plus post-dose paired global assessment; Test type: Superiority or Other; p = 1.0000, Wilcoxon signed-rank test
Statistical Analysis 3: Comparison: MultiHance 0.1 mmol/kg Arm (Reader 2); [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p < 0.0001, Wilcoxon signed-rank test
Statistical Analysis 4: Comparison: MultiHance 0.05 mmol/kg Arm (Reader 2); Null hypotheses: A 0.05 mmol/kg dose of MULTIHANCE is equal to a 0.1 mmol/kg dose of DOTAREM, in terms of the assessment of Extent of Disease in an off-site pre-dose plus postdose paired global assessment; Test type: Superiority or Other; p = 1.0000, Wilcoxon signed-rank test
Statistical Analysis 5: Comparison: MultiHance 0.1 mmol/kg Arm (Reader 3); [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.0023, Wilcoxon signed-rank test
Statistical Analysis 6: Comparison: MultiHance 0.05 mmol/kg Arm (Reader 3); [analysis description as in outcome 4, analysis 4]; Test type: Superiority or Other; p = 1.0000, Wilcoxon signed-rank test

5. Secondary Outcome: Lesion Contrast Enhancement
Description: as for outcome 1
Time Frame: Comparison of image sets obtained within 2 to 14 days
Measure: Number; unit: Participant Exams
Arm/Group | MultiHance 0.1 mmol/kg Arm (Reader 1) | MultiHance 0.1 mmol/kg Arm (Reader 2) | MultiHance 0.1 mmol/kg Arm (Reader 3) | MultiHance 0.05 mmol/kg Arm (Reader 1) | MultiHance 0.05 mmol/kg Arm (Reader 2) | MultiHance 0.05 mmol/kg Arm (Reader 3)
Number analyzed (Participants) | 63 | 62 | 62 | 96 | 94 | 95
Participant Exams
  MultiHance Better | 31 | 51 | 43 | 10 | 18 | 14
  No Difference between MultiHance and Dotarem | 31 | 9 | 17 | 77 | 56 | 64
  Dotarem Better | 1 | 2 | 2 | 9 | 20 | 17
Statistical Analysis 1: Comparison: MultiHance 0.1 mmol/kg Arm (Reader 1); Null hypotheses: A 0.1 mmol/kg dose of MULTIHANCE is equal to a 0.1 mmol/kg dose of DOTAREM, in terms of the assessment of Lesion Contrast Enhancement in an off-site pre-dose plus postdose paired global assessment; Test type: Superiority or Other; p < 0.0001, Wilcoxon signed-rank test
Statistical Analysis 2: Comparison: MultiHance 0.05 mmol/kg Arm (Reader 1); Null hypotheses: A 0.05 mmol/kg dose of MULTIHANCE is equal to a 0.1 mmol/kg dose of DOTAREM, in terms of the assessment of Lesion Contrast Enhancement in an off-site pre-dose plus post-dose paired global assessment; Test type: Superiority or Other; p = 1.0000, Wilcoxon signed-rank test
Statistical Analysis 3: Comparison: MultiHance 0.1 mmol/kg Arm (Reader 2); [analysis description as in outcome 5, analysis 1]; Test type: Superiority or Other; p < 0.0001, Wilcoxon signed-rank test
Statistical Analysis 4: Comparison: MultiHance 0.05 mmol/kg Arm (Reader 2); Null hypotheses: A 0.05 mmol/kg dose of MULTIHANCE is equal to a 0.1 mmol/kg dose of DOTAREM, in terms of the assessment of Lesion Contrast Enhancement in an off-site pre-dose plus postdose paired global assessment; Test type: Superiority or Other; p = 0.7503, Wilcoxon signed-rank test
Statistical Analysis 5: Comparison: MultiHance 0.1 mmol/kg Arm (Reader 3); [analysis description as in outcome 5, analysis 1]; Test type: Superiority or Other; p < 0.0001, Wilcoxon signed-rank test
Statistical Analysis 6: Comparison: MultiHance 0.05 mmol/kg Arm (Reader 3); Null hypotheses: A 0.05 mmol/kg dose of MULTIHANCE is equal to a 0.05 mmol/kg dose of DOTAREM, in terms of the assessment of Lesion Contrast Enhancement in an off-site pre-dose plus postdose paired global assessment; Test type: Superiority or Other; p = 0.5983, Wilcoxon signed-rank test

6. Secondary Outcome: Lesion to Background Ratio on Post T1-weighed Spin Echo Images
Description: The Unit of Measure is lesion-to-background ratio based on lesions assessed. For each lesion, Lesion-to-background ratio (LBR) = SI of lesion/SI of brain. Firstly, LBR of each lesion was assessed for each contrast agent postdose image separately, then the difference in LBR between MultiHance and Dotarem was calculated. The number presented in the result table below is "the mean difference in LBR postdose (MultiHance - Dotarem)"
Time Frame: 5-10 minutes Postdose
Measure: Mean (Standard Deviation); unit: ratio based on lesions assessed
Units Other Than Participants: Lesions
Arm/Group | MultiHance 0.1 mmol/kg Arm (Reader 1) | MultiHance 0.1 mmol/kg Arm (Reader 2) | MultiHance 0.1 mmol/kg Arm (Reader 3) | MultiHance 0.05 mmol/kg Arm (Reader 1) | MultiHance 0.05 mmol/kg Arm (Reader 2) | MultiHance 0.05 mmol/kg Arm (Reader 3)
Number analyzed (Participants) | 63 | 62 | 62 | 96 | 94 | 95
Number analyzed (Lesions) | 64 | 66 | 54 | 85 | 89 | 78
ratio based on lesions assessed | 0.22 (0.24) | 0.24 (0.20) | 0.21 (0.23) | -0.01 (0.21) | 0.03 (0.15) | 0.01 (0.15)
Statistical Analysis 1: Comparison: MultiHance 0.1 mmol/kg Arm (Reader 1); Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Mixed effect model with period, sequence, and IP and fixed effect and subject nested within sequence as random effect
Statistical Analysis 2: Comparison: MultiHance 0.05 mmol/kg Arm (Reader 1); Test type: Superiority or Other; p = 0.6898, Mixed Models Analysis; Mixed effect model with period, sequence, and IP and fixed effect and subject nested within sequence as random effect
Statistical Analysis 3: Comparison: MultiHance 0.1 mmol/kg Arm (Reader 2); Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Mixed effect model with period, sequence, and IP and fixed effect and subject nested within sequence as random effect
Statistical Analysis 4: Comparison: MultiHance 0.05 mmol/kg Arm (Reader 2); Test type: Superiority or Other; p = 0.1156, Mixed Models Analysis; Mixed effect model with period, sequence, and IP and fixed effect and subject nested within sequence as random effect
Statistical Analysis 5: Comparison: MultiHance 0.1 mmol/kg Arm (Reader 3); Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis
Statistical Analysis 6: Comparison: MultiHance 0.05 mmol/kg Arm (Reader 3); Test type: Superiority or Other; p = 0.7726, Mixed Models Analysis

7. Secondary Outcome: Lesion-brain Contrast-to-noise Ratio
Description: The Unit of Measure is contrast-to-noise ratio based on lesions assessed. For each lesion, Lesion-brain Contrast-to-noise Ratio (CNR) = [(SI of lesion - SI of brain)/SD for SI of noise] on Postdose Images of each lesion was calculated for each contrast agent image separately, then the difference in CNR between MultiHance and Dotarem was calculated. The number presented in the result table below is "the mean difference in CNR (MultiHance - Dotarem)"
Time Frame: 5-10 minutes Postdose
Measure: Mean (Standard Deviation); unit: ratio based on lesions assessed
Units Other Than Participants: Lesions
Arm/Group | MultiHance 0.1 mmol/kg Arm (Reader 1) | MultiHance 0.1 mmol/kg Arm (Reader 2) | MultiHance 0.1 mmol/kg Arm (Reader 3) | MultiHance 0.05 mmol/kg Arm (Reader 1) | MultiHance 0.05 mmol/kg Arm (Reader 2) | MultiHance 0.05 mmol/kg Arm (Reader 3)
Number analyzed (Participants) | 63 | 62 | 62 | 96 | 94 | 95
Number analyzed (Lesions) | 64 | 66 | 54 | 85 | 89 | 78
ratio based on lesions assessed | 17.40 (36.14) | 31.82 (45.28) | 39.73 (65.26) | 15.72 (36.05) | 19.06 (29.37) | 23.03 (49.53)
Statistical Analysis 1: Comparison: MultiHance 0.1 mmol/kg Arm (Reader 1); Test type: Superiority or Other; p = 0.0002, Mixed Models Analysis; Investigation product (IP) effect from mixed model with period, sequence, and IP as fixed effects and subject nested within sequence as random effect
Statistical Analysis 2: Comparison: MultiHance 0.05 mmol/kg Arm (Reader 1); Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 7, analysis 1]
Statistical Analysis 3: Comparison: MultiHance 0.1 mmol/kg Arm (Reader 2); Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 7, analysis 1]
Statistical Analysis 4: Comparison: MultiHance 0.05 mmol/kg Arm (Reader 2); Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 7, analysis 1]
Statistical Analysis 5: Comparison: MultiHance 0.1 mmol/kg Arm (Reader 3); Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 7, analysis 1]
Statistical Analysis 6: Comparison: MultiHance 0.05 mmol/kg Arm (Reader 3); Test type: Superiority or Other; p = 0.0003, Mixed Models Analysis; [statistical method as in outcome 7, analysis 1]

ADVERSE EVENTS:
Time Frame: Up to 24 hours after contrast media injection
Description: All adverse events collected were categorized using MedDRA 17.1 and tabulated
Groups:
- Study Arm 1 / MultiHance 0.1 mmol/kg: Study Arm 1: MultiHance 0.1 mmol/kg/ Experienced after dosed with MultiHance 0.1 mmol/kg.
  31 (MH as 1st injection) + 34 (MH as 2nd injection) = 65
- Study Arm 1 / Dotarem 0.1 mmol/kg: Study Arm 1: MultiHance 0.1 mmol/kg/ Experienced after dosed with Dotarem 0.1 mmol/kg.
  39 (Dotarem as 1st injection) + 31 (Dotarem as 2nd injection) =70
- Study Arm 2/ MultiHance 0.05 mmol/kg: Study Arm 2: MultiHance 0.05 mmol/kg/ Experienced after dosed with MultiHance 0.05 mmol/kg.
  53 (MH as 1st injection) + 51 (MH as 2nd injection) = 104
- Study Arm 2 / Dotarem 0.1 mmol/kg: Study Arm 2: MultiHance 0.05 mmol/kg/ Experienced after dosed with Dotarem 0.1 mmol/kg.
  54 (Dotarem as 1st injection) + 51 (Dotarem as 2nd injection) =105
Arm/Group | Study Arm 1 / MultiHance 0.1 mmol/kg | Study Arm 1 / Dotarem 0.1 mmol/kg | Study Arm 2/ MultiHance 0.05 mmol/kg | Study Arm 2 / Dotarem 0.1 mmol/kg
Serious Adverse Events (participants affected / at risk) | 0/65 | 0/70 | 0/104 | 0/105
Other Adverse Events (participants affected / at risk) | 1/65 | 2/70 | 3/104 | 7/105
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Study Arm 1 / MultiHance 0.1 mmol/kg (N=65) | Study Arm 1 / Dotarem 0.1 mmol/kg (N=70) | Study Arm 2/ MultiHance 0.05 mmol/kg (N=104) | Study Arm 2 / Dotarem 0.1 mmol/kg (N=105)
Skin infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0) | 2 (2)
Injection site swelling (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Injection site pruritus (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Procedural pain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dysgeusia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Study results may be presented at scientific symposia or published in a peer-review journal after review by sponsor in accordance with the guidelines set forth in the applicable publication or financial agreement